CLINICAL TRIAL: NCT04588298
Title: A Randomised, Open-Label, Parallel-Group, Pre-surgical Study to Investigate the Biological Effects of AZD9833 in Women With ER-positive, HER2-negative Primary Breast Cancer (SERENA-3)
Brief Title: A Study to Investigate the Biological Effects of AZD9833 in Women With ER-positive, HER2 Negative Primary Breast Cancer
Acronym: SERENA-3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8530C00003; 2020-001079-33 (EudraCT Number)
Record Dates: First submitted 2020-09-08; First posted 2020-10-19 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: HER2-negative Breast Cancer
Keywords: Breast cancer; Breast carcinoma; Estrogen-Receptor-positive breast cancer; HER2-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — AZD9833

STUDY DESIGN:
Intervention Model Description: This is a randomised, open-label, parallel-group study. The study is divided into three stages as follows:
  1. Stage 1: In this stage post-menopausal participants will be randomised in 2 cohorts in 1:1 ratio to receive AZD9833 with 12 evaluable participants in each cohort.
  2. Stage 2: In this stage post-menopausal participants may be randomised in up to 3 cohorts, which may include up to 3 doses of AZD9833.
  3. Stage 3 : In this stage post-menopausal participants may be randomised in up to 2 cohorts in 1:1 ratio, which may include up to 2 doses of AZD9833.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Stage 1: AZD9833 Dose A (Experimental): Post-menopausal participants will receive once daily oral dose A of AZD9833 in stage 1 of the study.
  Interventions: Drug: AZD9833
- Stage 1: AZD9833 Dose B (Experimental): Post-menopausal participants will receive once daily oral dose B of AZD9833 in stage 1 of the study.
  Interventions: Drug: AZD9833
- Stage 2: AZD9833 Dose A (Experimental): Post-menopausal participants will receive once daily oral dose A of AZD9833 in stage 2 of the study.
  Interventions: Drug: AZD9833
- Stage 2: AZD9833 Dose B (Experimental): Post-menopausal participants will receive once daily oral dose B of AZD9833 in stage 2 of the study.
  Interventions: Drug: AZD9833
- Stage 2: AZD9833 Dose C (Experimental): Post-menopausal participants will receive once daily oral dose C of AZD9833 in stage 2 of the study.
  Interventions: Drug: AZD9833
- Stage 3: AZD9833 Dose A (Experimental): Post-menopausal participants will receive once daily oral dose A of AZD9833 in stage 3 of the study.
  Interventions: Drug: AZD9833
- Stage 3: AZD9833: Dose B (Experimental): Post-menopausal participants will receive once daily oral dose B of AZD9833 in stage 3 of the study.
  Interventions: Drug: AZD9833

INTERVENTIONS:
Drug: AZD9833 — AZD9833 tablets will be administered orally.

SUMMARY:
This is a randomised, open-label, parallel-group, pre-surgical study aimed to investigate the biological effects, safety, tolerability, and pharmacokinetics (PK) of different doses of oral AZD9833 in post-menopausal women with primary breast cancer

DETAILED DESCRIPTION:
The study will be conducted in approximately 20 study centers across 3 countries and will be conducted in three stages (stage 1, stage 2 and stage 3). After the screening visit and confirmation of eligibility, evaluable participants will be enrolled across treatment groups. In stage 1, up to 24 evaluable participants across two treatment groups will be enrolled. A Safety and Data Monitoring Committee will convene to review stage 1 data and decide whether further treatment groups are required in stage 2. Stage 2 will include participants across up to 3 treatment groups. Stage 3 will include two treatment groups:

Stage 1 Group 1: AZD9833 Dose A once daily Group 2: AZD9833 Dose B once daily

Stage 2 Group 1: AZD9833 Dose A once daily Group 2: AZD9833 Dose B once daily Group 3: AZD9833 Dose C once daily

Stage 3 Group 1: AZD9833 Dose A once daily Group 2: AZD9833 Dose B once daily

Adverse events and concomitant medications information will be collected throughout the study. Thereafter there will be 28-day follow-up visit after discontinuation of study treatment

ELIGIBILITY:
Inclusion criteria:

* Provision of written informed consent prior to study entry
* Female participants aged at least 18 years
* Post-menopausal status defined as meeting at least one of the following criteria:

  1. Have undergone a bilateral oophorectomy
  2. Age ≥ 60 years
  3. Age ≥ 50 and < 60 years and with cessation of menses ≥ 12 months and follicle-stimulating hormone and oestradiol levels in the post-menopausal range and with an intact uterus in the absence of oral contraception or hormone replacement therapy prior to the diagnosis of breast cancer
* Female participants with newly diagnosed primary breast cancer scheduled to undergo treatment with curative intent by surgery and irrespective of clinical node status
* Histologically confirmed invasive breast cancer involving a palpable tumour of any size, or a tumour with an ultrasound assessed diameter of ≥ 1.0 cm
* Participants with adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 3 months can be considered for the study
* According to the local laboratory participants must have:

  1. ER positive breast cancer
  2. HER2-negative breast cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1

Exclusion Criteria:

* Previous systemic or local treatment for the new primary breast cancer currently under investigation (including surgery, radiotherapy, cytotoxic and endocrine treatments)
* Intervention with any of the following:

  1. Use of sex-hormone-containing drugs within 6 months prior to the first dose of study treatment
  2. Medications or herbal supplements known to be strong inhibitors/inducers of CYP3A4/5, sensitive CYP2B6 substrates and drugs which are substrates of CYP2C9 and/or CYP2C19 which have a narrow therapeutic index
  3. Drugs that are known to prolong QT and have a known risk of torsades de pointes
* Inflammatory breast cancer
* Any evidence of severe or uncontrolled systemic diseases which in the investigator's opinion makes it undesirable for the participant to participate in the study
* Any of the following cardiovascular criteria: Mean resting QTcF > 470 msec; resting heart rate of < 50 bpm for stages 1 and 2 at screening;resting heart rate <60 bpm at screening for Stage 3; any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG; any factors that increase the risk of QTc prolongation or risk of arrhythmic events; known left ventricular ejection fraction < 50%; significant cardiovascular procedure or event within the last 6 months; uncontrolled hypertension or symptomatic hypotension
* Inadequate bone marrow reserve or organ function
* Refractory nausea and vomiting, uncontrolled chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of AZD9833
* History of hypersensitivity to active or inactive excipients of AZD9833
* Previous randomisation in the present study
* Judgement by the Investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 135 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Robertson, Principal Investigator — Graduate Entry Medicine & Health School, University of Nottingham, Royal Derby Hospital
Locations (9):
- Georgia (2):
  - Research Site, Batumi
  - Research Site, Tbilisi
- Mexico (2):
  - Research Site, Aguascalientes
  - Research Site, Mexico City
- United Kingdom (5):
  - Research Site, Derby
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Hamilton E, Oliveira M, Turner N, Garcia-Corbacho J, Hernando C, Ciruelos EM, Kabos P, Ruiz-Borrego M, Armstrong A, Patel MR, Vaklavas C, Twelves C, Boni V, Incorvati J, Brier T, Gibbons L, Klinowska T, Lindemann JPO, Morrow CJ, Sykes A, Baird RD. A phase I dose escalation and expansion trial of the next-generation oral SERD camizestrant in women with ER-positive, HER2-negative advanced breast cancer: SERENA-1 monotherapy results. Ann Oncol. 2024 Aug;35(8):707-717. doi: 10.1016/j.annonc.2024.04.012. Epub 2024 May 8. PMID 38729567
- See also: BreastCancerStudyLocator.com — https://breastcancerstudylocator.com/
- See also: CSP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8530C00003&attachmentIdentifier=b92438e0-a17d-48e2-9fa2-230ec6b82e6f&fileName=AZ_D8530C00003_(PXL_247887)_CSP_final_Redacted.pdf&versionIdentifier=
- See also: SAP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8530C00003&attachmentIdentifier=2345d4d0-4f30-4d98-af8f-11f6537acafb&fileName=AZ_D8530C00003_(PXL_247887)_SAP_final_Redacted.pdf&versionIdentifier=
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8530C00003&attachmentIdentifier=8a4daf67-edac-43a7-b0ce-b4dd3d4c7abd&fileName=AZ_D8530C00003_(PXL_247887)_CSR_Synopsis_final_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 13 sites in 3 countries between November 2, 2020 and June 19, 2023.
Pre-assignment Details: Patients were enrolled according to the inclusion/exclusion criteria, with a 21 day screening period. Assessments were performed as per schedule. The study consists of 3 stages with different patients in each stage. Results pool data from the 75mg and 150mg arms of stages 1 and 2. This is per the predefined statistical analysis plan, which describes the combination of identical treatments in terms of dose and treatment duration. Stage 3 explored a different duration so is reported separately.
Groups:
- AZD9833 75 mg (Stage 1 + 2): Patients received once daily oral dose of AZD9833 75 mg for 5 to 7 days, during the study.
- AZD9833 150 mg (Stage 1 + 2): Patients received once daily oral dose of AZD9833 150 mg for 5 to 7 days, during the study.
- AZD9833 300 mg (Stage 2): Patients received once daily oral dose of AZD9833 300 mg for 5 to 7 days , during the study
- AZD9833 75 mg (Stage 3): Patients received once daily oral dose of AZD9833 75 mg for 12 to 15 days , during the study
- AZD9833 150 mg (Stage 3): Patients received once daily oral dose of AZD9833 150 mg for 12 to 15 days , during the study
Period: Overall Study
Arm/Group | AZD9833 75 mg (Stage 1 + 2) | AZD9833 150 mg (Stage 1 + 2) | AZD9833 300 mg (Stage 2) | AZD9833 75 mg (Stage 3) | AZD9833 150 mg (Stage 3)
Started | 30 | 33 | 13 | 30 | 29
Completed | 29 | 33 | 12 | 29 | 27
Not Completed | 1 | 0 | 1 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set was defined as all patients who received any amount of study treatment, regardless of whether that was the randomized therapy intended.
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD9833 75 mg (Stage 1 + 2) | AZD9833 150 mg (Stage 1 + 2) | AZD9833 300 mg (Stage 2) | AZD9833 75 mg (Stage 3) | AZD9833 150 mg (Stage 3) | Total
Number analyzed (Participants) | 30 | 33 | 13 | 30 | 29 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Mean and S.D data for Stage 1, and 2 combined, and stage 2, and stage 3 have been presented in 2 different rows.
  Years | 62.0 (7.35) | 65.7 (7.53) | 66.3 (8.20) | 64.0 (8.65) | 67.2 (10.03) | 64.9 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 33 | 13 | 30 | 29 | 135
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 30 | 33 | 13 | 30 | 29 | 135
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 4 | 5 | 9
  Not Hispanic or Latino | 29 | 32 | 13 | 26 | 24 | 124
  Other | 1 | 1 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Estrogen Receptor (ER) Expression Between Pre- and On-treatment Tumour Samples (Primary Analysis)
Description: The pharmacodynamic (PD) effect of AZD9833 on ER expression comparing pre- and on-treatment tumour samples in women with early breast cancer after 5 to 7 days and 12 to 15 days of AZD9833 treatment was assessed. The assessment was done by immunohistochemistry (IHC) method. The percentage change was calculated from an analysis of covariance (ANCVOA) model adjusting for baseline ER score and day of on-treatment biopsy.
Time Frame: Baseline (Screening Day -21 to 1) to Biopsy day (Days 5-7 [Stage 1 and 2] or Days 12-15 [Stage 3])
Population: PD analysis set included: all the patient who had taken at least 5 consecutive daily doses (Stage 1 and 2) or at least 12 consecutive daily doses (Stage 3) of AZD9833. The patient received last AZD9833 dose within 12 hours of the on-treatment biopsy, diagnostic and on-treatment biopsy pair was considered evaluable by central pathology assessment (>100 tumor cells per FFPE biopsy, and minimum of 2 slides for ER measurement), with no protocol deviations affecting the biomarker analysis.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage change from baseline
Arm/Group | AZD9833 75 mg (Stage 1 + 2) | AZD9833 150 mg (Stage 1 + 2) | AZD9833 300 mg (Stage 2) | AZD9833 75 mg (Stage 3) | AZD9833 150 mg (Stage 3)
Number analyzed (Participants) | 26 | 31 | 11 | 24 | 26
Percentage change from baseline | -62.7 [-67.46 to -57.93] | -62.8 [-67.13 to -58.43] | -67.1 [-74.49 to -59.74] | -66.9 [-72.34 to -61.46] | -65.0 [-70.27 to -59.81]

2. Primary Outcome: Percentage Change From Baseline in ER Expression Between Pre- and On-treatment Tumour Samples (Sensitivity Analysis)
Description: The PD effect of AZD9833 on ER expression comparing pre- and on-treatment tumour samples in women with early breast cancer after 5 to 7 days and 12 to 15 days of AZD9833 treatment was assessed. The assessment was done by IHC method. The sensitivity analysis excluded any patients who were HER2-positive patient by central assessment as well as patients with baseline ER H-score < 10. The percentage change was calculated from ANCVOA model adjusting for baseline ER score and day of on-treatment biopsy.
Time Frame: Baseline (Screening Day -21 to 1) to Biopsy Day (Days 5-7 [Stage 1 and 2] or Days 12-15 [Stage 3])
Population: as for outcome 1
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage change from baseline
Arm/Group | AZD9833 75 mg (Stage 1 + 2) | AZD9833 150 mg (Stage 1 + 2) | AZD9833 300 mg (Stage 2) | AZD9833 75 mg (Stage 3) | AZD9833 150 mg (Stage 3)
Number analyzed (Participants) | 25 | 31 | 11 | 24 | 26
Percentage change from baseline | -62.1 [-67.00 to -57.25] | -62.3 [-66.64 to -57.88] | -66.6 [-74.00 to -59.14] | -66.9 [-72.34 to -61.46] | -65.0 [-70.27 to -59.81]

3. Secondary Outcome: Percentage Change From Baseline in Progesterone Receptor (PgR) Expression Between Pre- and On-treatment Tumour Samples (Primary Analysis)
Description: The PD effects of AZD9833 on PgR expression comparing pre- and on-treatment tumour samples in women with early breast cancer after 5 to 7 days and 12 to 15 days of AZD9833 treatment was assessed. The assessment was done by IHC method. The percentage change was calculated from an ANCOVA model adjusting for baseline PgR score and day of on-treatment biopsy.
Time Frame: Baseline (Screening Day -21 to 1) to Biopsy Day (Days 5-7 [Stage 1 and 2] or Days 12-15 [Stage 3])
Population: PD analysis set included: all the patient who had taken at least 5 consecutive daily doses (Stage 1 and 2) or at least 12 consecutive daily doses (Stage 3) of AZD9833. The patient received last AZD9833 dose within 12 hours of the on-treatment biopsy, diagnostic and on-treatment biopsy pair was considered evaluable by central pathology assessment (>100 tumor cells per FFPE biopsy, and minimum of 2 slides for PgR measurement), with no protocol deviations affecting the biomarker analysis.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage change from baseline
Arm/Group | AZD9833 75 mg (Stage 1 + 2) | AZD9833 150 mg (Stage 1 + 2) | AZD9833 300 mg (Stage 2) | AZD9833 75 mg (Stage 3) | AZD9833 150 mg (Stage 3)
Number analyzed (Participants) | 26 | 31 | 11 | 24 | 26
Percentage change from baseline | 194.8 [25.50 to 364.03] | -3.0 [-158.37 to 152.36] | 170.3 [-89.67 to 430.33] | -24.2 [-547.03 to 498.69] | 463.8 [-38.45 to 966.02]

4. Secondary Outcome: Percentage Change From Baseline in PgR Expression Between Pre- and On-treatment Tumour Samples (Sensitivity Analysis)
Description: The PD effects of AZD9833 on PgR expression comparing pre- and on-treatment tumour samples in women with early breast cancer after 5 to 7 days and 12 to 15 days of AZD9833 treatment was assessed. The assessment was done by IHC method. The sensitivity analysis excluded any patients who were HER2-positive patient by central assessment as well as patients with baseline PgR H-score < 10. The percentage change was calculated from an ANCOVA model adjusting for baseline PgR score and day of on-treatment biopsy.
Time Frame: Baseline (Screening Day -21 to 1) to Biopsy day (Days 5-7 [Stage 1 and 2] or Days 12-15 [Stage 3])
Population: as for outcome 3
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage change from baseline
Arm/Group | AZD9833 75 mg (Stage 1 + 2) | AZD9833 150 mg (Stage 1 + 2) | AZD9833 300 mg (Stage 2) | AZD9833 75 mg (Stage 3) | AZD9833 150 mg (Stage 3)
Number analyzed (Participants) | 19 | 26 | 8 | 23 | 20
Percentage change from baseline | -35.2 [-45.86 to -24.57] | -44.0 [-53.09 to -34.90] | -36.7 [-52.96 to -20.52] | -61.8 [-76.93 to -46.62] | -55.0 [-71.29 to -38.78]

5. Secondary Outcome: Percentage Change From Baseline in Ki-67 Labelling Index Between Pre- and On-treatment Tumour Samples (Primary Analysis)
Description: The PD effect of AZD9833 on antigen Ki-67 expression comparing pre- and on-treatment tumour samples in women with early breast cancer after 5 to 7 days and 12 to 15 days of AZD9833 treatment was assessed. The assessment was done by IHC method. The percentage change was calculated from an ANCOVA model adjusting for log baseline Ki67 index and day of on-treatment biopsy. The Ki-67 index data were log transformed prior to analysis, with results back-transformed to represent percentage change.
Time Frame: Baseline (Screening Day -21 to 1) to Biopsy day (Days 5-7 [Stage 1 and 2] or Days 12-15 [Stage 3])
Population: PD analysis set included: all the patient who had taken at least 5 consecutive daily doses (Stage 1 and 2) or at least 12 consecutive daily doses (Stage 3) of AZD9833. The patient received last AZD9833 dose within 12 hours of the on-treatment biopsy, diagnostic and on-treatment biopsy pair was considered evaluable by central pathology assessment (>100 tumor cells per FFPE biopsy, and minimum of 2 slides for Ki-67 measurement), with no protocol deviations affecting the biomarker analysis.
Measure: Geometric Least Squares Mean (80% Confidence Interval); unit: Percentage change from baseline
Arm/Group | AZD9833 75 mg (Stage 1 + 2) | AZD9833 150 mg (Stage 1 + 2) | AZD9833 300 mg (Stage 2) | AZD9833 75 mg (Stage 3) | AZD9833 150 mg (Stage 3)
Number analyzed (Participants) | 26 | 31 | 11 | 24 | 26
Percentage change from baseline | -40.3 [-52.78 to -24.49] | -79.4 [-83.37 to -74.55] | -78.2 [-84.82 to -68.77] | -73.0 [-79.42 to -64.64] | -77.5 [-82.68 to -70.86]

6. Secondary Outcome: Percentage Change From Baseline in Ki-67 Labelling Index Between Pre- and On-treatment Tumour Samples (Sensitivity Analysis)
Description: The PD effect of AZD9833 on antigen Ki-67 expression comparing pre- and on-treatment tumour samples in women with early breast cancer after 5 to 7 days and 12 to 15 days of AZD9833 treatment was assessed. The assessment was done by IHC method. The sensitivity analysis excluded any patients who were HER2-positive patient by central assessment as well as patients with baseline Ki67 labelling index <5%. The percentage change was calculated from an ANCOVA model adjusting for log baseline Ki67 index and day of on-treatment biopsy. The Ki-67 index data were log transformed prior to analysis, with results back-transformed to represent percentage change.
Time Frame: Baseline (Screening Day -21 to 1) to Biopsy Day (Days 5-7 [Stage 1 and 2] or Days 12-15 [Stage 3])
Population: as for outcome 5
Measure: Geometric Least Squares Mean (80% Confidence Interval); unit: Percentage change from baseline
Arm/Group | AZD9833 75 mg (Stage 1 + 2) | AZD9833 150 mg (Stage 1 + 2) | AZD9833 300 mg (Stage 2) | AZD9833 75 mg (Stage 3) | AZD9833 150 mg (Stage 3)
Number analyzed (Participants) | 17 | 28 | 11 | 18 | 20
Percentage change from baseline | -49.3 [-62.18 to -31.96] | -81.3 [-85.14 to -76.49] | -78.9 [-85.37 to -69.46] | -81.7 [-86.45 to -75.24] | -81.9 [-86.38 to -75.88]

7. Secondary Outcome: Number of Patients With Adverse Events (AEs)
Description: The safety and tolerability of AZD9833 in this patient population was evaluated.
Time Frame: From screening (Day -21 to 1) through 28-day follow-up (Upto 2 months)
Population: Safety Analysis Set is defined as all patients who received any amount of study treatment, regardless of whether that was the randomized therapy at intended.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD9833 75 mg (Stage 1 + 2) | AZD9833 150 mg (Stage 1 + 2) | AZD9833 300 mg (Stage 2) | AZD9833 75 mg (Stage 3) | AZD9833 150 mg (Stage 3)
Number analyzed (Participants) | 30 | 33 | 13 | 30 | 29
Participants
  Any AE | 9 | 17 | 9 | 11 | 19
  Any AE possibly related to treatment | 4 | 14 | 6 | 10 | 17
  Any AE of CTCAE grade 3 or higher | 0 | 1 | 0 | 0 | 0
  Any AE of CTCAE grade 3 or higher, possibly related to treatment | 0 | 1 | 0 | 0 | 0
  Any AE with outcome = death | 0 | 0 | 0 | 0 | 0
  Any AE with outcome = death, possibly related to treatment | 0 | 0 | 0 | 0 | 0
  Any SAE (including events with outcome = death) | 0 | 0 | 0 | 0 | 0
  Any SAE (including events with outcome = death), possibly related to treatment | 0 | 0 | 0 | 0 | 0
  Any SAE leading to discontinuation of treatment | 0 | 0 | 0 | 0 | 0
  Any SAE leading to discontinuation of treatment, possibly related to treatment | 0 | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of treatment | 0 | 0 | 1 | 0 | 2
  Any AE leading to discontinuation of treatment, possibly related to treatment | 0 | 0 | 0 | 0 | 2
  Any AE leading to dose modification of treatment | 0 | 0 | 0 | 0 | 0
  Any AE leading to dose modification of treatment, possibly related to treatment | 0 | 0 | 0 | 0 | 0
  Any other significant AEs | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Plasma Concentrations of AZD9833
Description: The plasma concentration of AZD9833 in this participant population was evaluated
Time Frame: Days 5-7 or Days 12-15 (Pre and Post biopsy)
Population: The Pharmacokinetic (PK) Analysis Set is defined as all patients who received at least one dose of AZD9833 per protocol, for whom there is at least one reportable PK concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | AZD9833 75 mg (Stage 1 + 2) | AZD9833 150 mg (Stage 1 + 2) | AZD9833 300 mg (Stage 2) | AZD9833 75 mg (Stage 3) | AZD9833 150 mg (Stage 3)
Number analyzed (Participants) | 29 | 33 | 12 | 28 | 27
Nanograms per milliliter
  Days 5-7 or Days 12-15 (Pre-biopsy): number analyzed (Participants) | 28 | 33 | 12 | 28 | 27
  Days 5-7 or Days 12-15 (Pre-biopsy) | 50.712 (74.1) | 122.134 (103.8) | 180.773 (173.3) | 46.939 (56.3) | 120.516 (70.0)
  Days 5-7 or Days 12-15 (Post-biopsy): number analyzed (Participants) | 29 | 32 | 12 | 28 | 27
  Days 5-7 or Days 12-15 (Post-biopsy) | 58.304 (62.2) | 142.916 (102.4) | 213.446 (175.6) | 54.075 (42.8) | 137.687 (55.4)

ADVERSE EVENTS:
Time Frame: From screening (Day -21 to 1) through 28-day follow-up (Up to 2 months)
Arm/Group | AZD9833 75 mg (Stage 1 + 2) | AZD9833 150 mg (Stage 1 + 2) | AZD9833 300 mg (Stage 2) | AZD9833 75 mg (Stage 3) | AZD9833 150 mg (Stage 3)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/33 | 0/13 | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/33 | 0/13 | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 7/30 | 17/33 | 9/13 | 11/30 | 19/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9833 75 mg (Stage 1 + 2) (N=30) | AZD9833 150 mg (Stage 1 + 2) (N=33) | AZD9833 300 mg (Stage 2) (N=13) | AZD9833 75 mg (Stage 3) (N=30) | AZD9833 150 mg (Stage 3) (N=29)
Visual impairment (Eye disorders) | 0 (0) | 5 (11) | 3 (6) | 6 (23) | 7 (10)
Photopsia (Eye disorders) | 2 (2) | 4 (6) | 2 (2) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 3 (4) | 1 (1) | 4 (5)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (4) | 1 (4) | 2 (2) | 1 (2)
Diplopia (Eye disorders) | 0 (0) | 4 (10) | 1 (1) | 0 (0) | 5 (8)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 3 (3)
Fatigue (General disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Vision blurred (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2022-07-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT04588298/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT04588298/SAP_001.pdf